CLINICAL TRIAL: NCT02201420
Title: Evaluation of Technetium Tc 99m Tilmanocept Localization, Retention, and Distribution in Primary Cutaneous Kaposi's Sarcoma (KS) and Lymphatic Drainage From KS Lesions by SPECT/CT Imaging.
Brief Title: Evaluation of Tc 99m Tilmanocept Localization in Primary Cutaneous Kaposi's Sarcoma and Lymphatic Drainage by SPECT/CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-12
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Kaposi's Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tc 99m tilmanocept (Experimental): Subjects who are enrolled and will receive 50 micrograms tilmanocept radiolabeled with 2 millicuries of Tc 99m and undergo serial SPECT or SPECT/CT imaging.
  Interventions: Drug: Tc 99m tilmanocept

INTERVENTIONS:
Drug: Tc 99m tilmanocept
  Other Names: Lymphoseek

SUMMARY:
The purpose of this study (NAV3-12) is to determine the dissemination and localization of Tc 99m tilmanocept by SPECT and SPECT/CT imaging in subjects with confirmed cutaneous KS. This is a single center, open-label, within-subject study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent with Health Insurance Portability and Accountability Act (HIPAA) authorization before the initiation of any study-related procedures.
2. The subject is at least 18 years of age at the time of consent.
3. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 to 2.
4. The subject has a KS stage of T(0), I(0), S(0).
5. The subject has a marker lesion with a confirmed diagnosis of KS (CD 206-expressing cutaneous KS) via punch biopsy. The location of the marker KS lesion will be limited to locations on the extremities: from the shoulder to the metacarpal region or from the groin to the metatarsal region.
6. The subject has a marker KS lesion that is ≥ 1cm in diameter.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has had prior chemotherapy, immunotherapy, or radiation therapy to the local KS site or regional lymphatic system within one year of enrollment.
3. The subject has undergone node basin surgery of any type or radiation to the nodal basin(s) potentially draining the marker KS lesion.
4. The subject has known sensitivity to dextran.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie C Abbruzzese, MS, RD, CCRA, Study Director — Navidea Biopharmaceuticals
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Tc 99m Tilmanocept: Subjects who are enrolled and will receive 50 micrograms tilmanocept radiolabeled with 2 millicuries of Tc 99m and undergo serial SPECT or SPECT/CT imaging.
  Tc 99m tilmanocept
Period: Overall Study
Arm/Group | Tc 99m Tilmanocept
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tc 99m Tilmanocept
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
HIV Diagnosis [Number; unit: participants]
  HIV+ | 4
  HIV- | 1

OUTCOME MEASURES:

1. Primary Outcome: Localization
Description: Count of subjects with a localization by Tc 99m tilmanocept by imaging. Localization is based on the use of SPECT imaging and defined as the accumulation of radioactivity at intensity greater than background.
Time Frame: Up to 4 days
Measure: Number; unit: participants
Arm/Group | Tc 99m Tilmanocept
Number analyzed (Participants) | 5
participants | 5

2. Secondary Outcome: Time to Localization
Description: Number of Participants with Localization at One Hour
Time Frame: 1 hour
Measure: Number; unit: participants localizing in 1 hour
Arm/Group | Tc 99m Tilmanocept
Number analyzed (Participants) | 5
participants localizing in 1 hour | 5

ADVERSE EVENTS:
Arm/Group | Tc 99m Tilmanocept
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tc 99m Tilmanocept (N=5)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Leg Edema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not submit a publication to journals or professional societies without the prior written approval of the Sponsor.